CLINICAL TRIAL: NCT07320235
Title: IMetelstat and Azacitidine With or Without Venetoclax GIveN in rElapsed Acute Myeloid Leukemia (IMAGINE Trial)
Brief Title: Imetelstat Combinations in Relapsed AML
Acronym: IMAGINE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Douglas Tremblay (Other)
Collaborators: Geron Corporation (Industry)
Responsible Party: Sponsor-Investigator, Douglas Tremblay, Associate Professor, Division of Hematology Oncology, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-25-01212; PRMC-25-108 (Other: TCI PRMC)
Record Dates: First submitted 2025-12-09; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Relapsed Acute Myeloid Leukemia
Keywords: IMAGINE Trial; Acute Myeloid Leukemia; AML; Relapsed Acute Myeloid Leukemia; Imetelstat; Imetelstat and Azacitidine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — imetelstat; GRN163L peptide; Azacitidine; venetoclax

STUDY DESIGN:
Intervention Model Description: The trial will consist of a safety run-in phase (Part A) employing a 3+3 design to monitor dose-limiting toxicities of imetelstat when administered in combination with a fixed dose of azacitidine. Part B will consist of a phase 1b trial employing a BOIN12 design to determine the optimal biological dose of imetelstat, starting at a lower dose level, in combination with azacitidine and venetoclax.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A Safety Run-In phase: Imetelstat in combination with Azacitidine (Active Comparator): Part A combination therapy:
  * Imetelstat will be administered on Day 1 of each 28-day cycle
  * Azacitidine once daily for Days 1 (+/- 1 day) through 7 (+/- 1 day) of each 28-day cycle.
  Interventions: Drug: Imetelstat; Drug: Azacitidine
- Part B Combination Therapy: Imetelstat in combination with Azacitidine with or without Venetoclax (Active Comparator): * Imetelstat will be administered on Day 1 of each 28-day cycle
  * Azacitidine once daily for Days 1 (+/- 1 day) through 7 (+/- 1 day) of each 28-day cycle.
  * Venetoclax once daily for Days 1 (+/- 1 day) through 14 (+/- 1 day) of each 28-day cycle.

INTERVENTIONS:
Drug: Imetelstat — Three 3 dose levels administered on Day 1 of each 28-day cycle for Safety Run-in Phase and optimal dose to be administered on Day 1 of each 28-day cycle
  Other Names: GRN163L
  Arms: Part A Safety Run-In phase: Imetelstat in combination with Azacitidine
Drug: Azacitidine — 75mg/m2 IV or subcutaneous (SQ) once daily for Days 1 (+/- 1 day) through 7 (+/- 1 day) of each 28-day cycle. Azacitidine can be administered locally as long as documentation of administration is provided to the study team.
  Arms: Part A Safety Run-In phase: Imetelstat in combination with Azacitidine
Drug: Venetoclax — Venetoclax 400mg oral once daily for Days 1 (+/- 1 day) through 14 (+/- 1 day) of each 28-day cycle.
  Venetoclax reduced dosey should be substituted if concomitant posaconazole, or if other concomitant strong CYP3A4 inhibitor (e.g. voriconazole) or 200mg for moderate CYP3A4 inhibitor (e.g. isavuconazole).
  For Cycle 1, participants will receive a venetoclax ramp-up dose on day 1, day 2, and days 3-14 of venetoclax,.
  If the participant is being treated with concomitant posaconazole, or other concomitant strong CYP3A4 inhibitor, or with a concomitant moderate CYP3A4 inhibitor or a pg-p inhibitor, participants will receive a lower ramp-up dose on day 1, day 2, and days 3-14 of venetoclax.

SUMMARY:
IMAGINE is a two-part trial to evaluate the safety and preliminary efficacy of imetelstat in combination with azacitidine with or without venetoclax in patients with relapsed or refractory AML. The trial will consist of a safety run-in phase (Part A) employing a 3+3 design to monitor dose-limiting toxicities of imetelstat when administered in combination with a fixed dose of azacitidine. Part B will consist of a phase 1b trial employing a BOIN12 design to determine the optimal biological dose of imetelstat, starting at a lower dose level, in combination with azacitidine and venetoclax. Total of up to 36 participants will be accrued over 54 months at Mount Sinai Hospital. Estimated duration of trial is 114 months including recruitment, screening, treatment, and follow-up.

ELIGIBILITY:
Inclusion Criteria In order to be eligible for participation in this trial,

* Participants must be ≥18 years of age at time of signing the Informed Consent Form (ICF).
* Participants must voluntarily sign an ICF.
* Participants must have WHO-confirmed non-APL AML who have not responded to or relapsed after at least one prior therapy and for whom no standard therapy that may provide clinical benefit is available.

  o Participants with isolated extramedullary disease (EMD), including leukemia cutis, are included but not those with active known CNS disease.
* Participants must have a life expectancy of at least 12 weeks per investigator.
* ECOG performance status ≤ 3.
* Women of child bearing potential (WOCBP), defined as a sexually mature woman not surgically sterilized or post-menopausal for at least 24 consecutive months if ≤55 years or 12 months if >55 years, must have a negative serum pregnancy test at screening and cycle 1 day 1 and must agree to use highly effective methods of birth control starting with the first dose of study therapy through 6 months after the last dose of study therapy. Highly effective methods of contraception include double-barrier methods (diaphragm with spermicidal gel and condoms with spermicide), partner vasectomy, and total abstinence
* Male participants should agree to use a highly effective method of contraception starting with the first dose of study therapy through 6 months after the last dose of study therapy. 8. Must have adequate organ function as demonstrated by the following:

  * Serum total bilirubin ≤ 2.0 x upper limit of normal (ULN) unless considered due to leukemic organ involvement or Gilbert's syndrome.
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN.
  * Creatinine clearance (CrCl) ≥ 30 mL/min (measured or estimated by Cockcroft-Gault formula).
* Ability to adhere to the study visit schedule and all protocol requirements.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria The participant must be excluded from participating in the trial if the participant:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 2 weeks or within 5 half-lives of the prior investigational agent, whichever is shorter, of the first dose of treatment.
* Known clinically active central nervous system (CNS) leukemia. a. Prior CNS leukemia will be allowed if the most recent cerebral spinal fluid sample is negative prior to study initiation and there is no clinical suspicion for active CNS disease.
* Has a white blood cell count > 25 x 109/L (hydroxyurea and/or continuous cytarabine ≤1 g/m2 is permitted to meet this criterion).
* Active Graft Versus Host Disease (GVHD), or any GVHD requiring treatment with immunosuppression, with the exception of topical steroids and systemic steroids at a dose equivalent to prednisone 10mg or less. Any GVHD treatment (including calcineurin inhibitors) must be discontinued at least 28 days prior to Day 1 of study treatment.
* Participants with a history of other cancers must not be receiving active treatment (with radiation or chemotherapy) and must be free of disease for 2 years prior to the Screening Visit with the exception of localized prostate cancer treated with hormone therapy, breast cancer treated with hormone therapy, localized basal cell carcinoma, non-melanoma skin cancer, cervical carcinoma in situ, concurrent low-grade lymphoma, that is asymptomatic and lacks bulky disease and shows no evidence of progression, and for which the participant is not receiving any systemic therapy or radiation
* Myocardial infarction or unstable angina within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.
* Presence of active serious infection. a. If a participant is identified to have COVID-19 during the screening period, participants may be considered eligible if in the opinion of the investigator there are no COVID-19 sequelae that may place the participant at a higher risk of receiving investigational treatment
* Any serious, unstable medical or psychiatric condition that would prevent, (as judged by the Investigator) the participant from signing the informed consent form or any condition, including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Known history of uncontrolled human immunodeficiency virus (HIV)
* Active known systemic hepatitis A, B, or C infection requiring therapy or known cirrhosis.
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is investigational site or pharmaceutical sponsor staff directly involved with this trial, unless prospective IRB approval (by chair or designee) is given allowing exception to this criterion for a specific participant.
* Organ transplant recipients other than bone marrow transplant.
* Women who are pregnant or lactating.
* Participants with known gastrointestinal (GI) disease or prior GI procedure that could interfere with the oral absorption or tolerance of venetoclax, including difficulty swallowing, are not eligible (Part B only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-06-17 (Estimated); Study Completion 2035-06-15 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Cycle 1 Day 1 up to Cycle 1 Day 28 (each cycle is 28 days), for 6 cycles
  The DLT-evaluable population includes participants in the Part A portion of the trial who received at least one dose of imetelstat and azacitidine and either experienced a Dose-Limiting Toxicity (DLT) during the first-cycle DLT assessment period or completed their first-cycle DLT assessment.

SECONDARY OUTCOMES:
Optimal Biological Dose (OBD) | Cycle 1 Day 1 up to Cycle 1 Day 28 (each cycle is 28 days), for 6 cycles
  The OBD-evaluable population includes participants in the Part B portion of the trial who received at least one dose of imetelstat, azacitidine, and venetoclax and either experienced a Dose-Limiting Toxicity (DLT) during the first-cycle DLT assessment period or completed their first-cycle DLT assessment.
  Optimal Biological Dose (OBD) is defined as the lowest safe dose providing the highest rate of efficacy.
Disease-Free Survival (DFS) | Cycle 1 Day 1 (each cycle is 28 days) until the first documented evidence of relapsed disease or death from any cause, or up to 6 months. whichever occurs first
  Disease-Free Survival (DFS) is defined as the time from the first occurrence of CR, CRh, or CRi, based on ELN 2022 response criteria (which, in this study, can only be assessed at cycles 2, 4, or 6), until the first documented evidence of relapsed disease or death from any cause, whichever occurs first.Participants who do not achieve CR, CRh, or CRi at one of their cycle 2, 4, or 6 assessments will be excluded from this analysis.
Duration of Response (DOR) | Cycle 1 Day 1 (each cycle is 28 days) until the first documented evidence of relapsed disease or death from any cause, or up to 6 months whichever occurs first
  Duration of Response (DOR) is defined as the time from the first occurrence of CR, CRh, CRi, MLFS, or PR based on ELN 2022 response criteria (which, in this study, can only be assessed at D22 of cycles 2, 4, or 6), until the first documented evidence of relapsed disease or death from any cause, whichever occurs first. Participants who do not achieve CR, CRh, Cri, MLFS, or PR at one of their cycle 2, 4, or 6 assessments will be excluded from this analysis.
Overall Survival (OS) | Cycle 1 Day 1 (each cycle is 28 days) to the date of death, regardless of the actual cause of death, or or up to 5 years, whichever comes first
  Overall Survival (OS) is defined as the time from C1D1 to the date of death, regardless of the actual cause of the participant's death. For participants who are still alive at the time of data analysis or who are lost to follow-up, OS time will be censored at the last recorded date that the participant is known to be alive as of the data cut-off date for the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Tremblay, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; John Mascarenhas, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD sharing plan is Undecided.

REFERENCES:
- [Background] Zeidan AM, Platzbecker U, Bewersdorf JP, Stahl M, Ades L, Borate U, Bowen D, Buckstein R, Brunner A, Carraway HE, Daver N, Diez-Campelo M, de Witte T, DeZern AE, Efficace F, Garcia-Manero G, Garcia JS, Germing U, Giagounidis A, Griffiths EA, Hasserjian RP, Hellstrom-Lindberg E, Iastrebner M, Komrokji R, Kulasekararaj AG, Malcovati L, Miyazaki Y, Odenike O, Santini V, Sanz G, Scheinberg P, Stauder R, van de Loosdrecht AA, Wei AH, Sekeres MA, Fenaux P. Consensus proposal for revised International Working Group 2023 response criteria for higher-risk myelodysplastic syndromes. Blood. 2023 Apr 27;141(17):2047-2061. doi: 10.1182/blood.2022018604. PMID 36724453
- [Background] Hayano RS, Adachi R. Estimation of the total population moving into and out of the 20 km evacuation zone during the Fukushima NPP accident as calculated using "Auto-GPS" mobile phone data. Proc Jpn Acad Ser B Phys Biol Sci. 2013;89(5):196-9. doi: 10.2183/pjab.89.196. PMID 23666090
- [Background] Antar AI, Otrock ZK, Jabbour E, Mohty M, Bazarbachi A. FLT3 inhibitors in acute myeloid leukemia: ten frequently asked questions. Leukemia. 2020 Mar;34(3):682-696. doi: 10.1038/s41375-019-0694-3. Epub 2020 Jan 9. PMID 31919472
- [Background] DiNardo CD, Wei AH. How I treat acute myeloid leukemia in the era of new drugs. Blood. 2020 Jan 9;135(2):85-96. doi: 10.1182/blood.2019001239. PMID 31765470
- [Background] DiNardo CD, Jonas BA, Pullarkat V, Thirman MJ, Garcia JS, Wei AH, Konopleva M, Dohner H, Letai A, Fenaux P, Koller E, Havelange V, Leber B, Esteve J, Wang J, Pejsa V, Hajek R, Porkka K, Illes A, Lavie D, Lemoli RM, Yamamoto K, Yoon SS, Jang JH, Yeh SP, Turgut M, Hong WJ, Zhou Y, Potluri J, Pratz KW. Azacitidine and Venetoclax in Previously Untreated Acute Myeloid Leukemia. N Engl J Med. 2020 Aug 13;383(7):617-629. doi: 10.1056/NEJMoa2012971. PMID 32786187
- [Background] Maiti A, Rausch CR, Cortes JE, Pemmaraju N, Daver NG, Ravandi F, Garcia-Manero G, Borthakur G, Naqvi K, Ohanian M, Short NJ, Alvarado Y, Kadia TM, Takahashi K, Yilmaz M, Jain N, Kornblau S, Montalban Bravo G, Sasaki K, Andreeff M, Bose P, Ferrajoli A, Issa GC, Jabbour EJ, Masarova L, Thompson PA, Wang S, Konoplev S, Pierce SA, Ning J, Qiao W, Welch JS, Kantarjian HM, DiNardo CD, Konopleva MY. Outcomes of relapsed or refractory acute myeloid leukemia after frontline hypomethylating agent and venetoclax regimens. Haematologica. 2021 Mar 1;106(3):894-898. doi: 10.3324/haematol.2020.252569. No abstract available. PMID 32499238
- [Background] Feld J, Tremblay D, Dougherty M, Czaplinska T, Sanchez G, Brady C, Kremyanskaya M, Bar-Natan M, Keyzner A, Marcellino BK, Gabrilove J, Navada SC, Silverman LR, El Jamal SM, Mascarenhas J, Shih AH. Safety and Efficacy: Clinical Experience of Venetoclax in Combination With Hypomethylating Agents in Both Newly Diagnosed and Relapsed/Refractory Advanced Myeloid Malignancies. Hemasphere. 2021 Mar 9;5(4):e549. doi: 10.1097/HS9.0000000000000549. eCollection 2021 Apr. PMID 33718803
- [Background] Pollyea DA, Bixby D, Perl A, Bhatt VR, Altman JK, Appelbaum FR, de Lima M, Fathi AT, Foran JM, Gojo I, Hall AC, Jacoby M, Lancet J, Mannis G, Marcucci G, Martin MG, Mims A, Neff J, Nejati R, Olin R, Percival ME, Prebet T, Przespolewski A, Rao D, Ravandi-Kashani F, Shami PJ, Stone RM, Strickland SA, Sweet K, Vachhani P, Wieduwilt M, Gregory KM, Ogba N, Tallman MS. NCCN Guidelines Insights: Acute Myeloid Leukemia, Version 2.2021. J Natl Compr Canc Netw. 2021 Jan 6;19(1):16-27. doi: 10.6004/jnccn.2021.0002. PMID 33406488
- [Background] HAYFLICK L, MOORHEAD PS. The serial cultivation of human diploid cell strains. Exp Cell Res. 1961 Dec;25:585-621. doi: 10.1016/0014-4827(61)90192-6. No abstract available. PMID 13905658
- [Background] Bodnar AG, Ouellette M, Frolkis M, Holt SE, Chiu CP, Morin GB, Harley CB, Shay JW, Lichtsteiner S, Wright WE. Extension of life-span by introduction of telomerase into normal human cells. Science. 1998 Jan 16;279(5349):349-52. doi: 10.1126/science.279.5349.349. PMID 9454332
- [Background] Harley CB, Futcher AB, Greider CW. Telomeres shorten during ageing of human fibroblasts. Nature. 1990 May 31;345(6274):458-60. doi: 10.1038/345458a0. PMID 2342578
- [Background] Diebold J, Raphael M, Prevot S, Audouin J. Lymphomas associated with HIV infection. Cancer Surv. 1997;30:263-93. PMID 9547997
- [Background] McEachern MJ, Krauskopf A, Blackburn EH. Telomeres and their control. Annu Rev Genet. 2000;34:331-358. doi: 10.1146/annurev.genet.34.1.331. PMID 11092831
- [Background] Harley CB. Telomerase is not an oncogene. Oncogene. 2002 Jan 21;21(4):494-502. doi: 10.1038/sj.onc.1205076. PMID 11850774
- [Background] Wright WE, Piatyszek MA, Rainey WE, Byrd W, Shay JW. Telomerase activity in human germline and embryonic tissues and cells. Dev Genet. 1996;18(2):173-9. doi: 10.1002/(SICI)1520-6408(1996)18:23.0.CO;2-3. PMID 8934879
- [Background] Chiu CP, Harley CB. Replicative senescence and cell immortality: the role of telomeres and telomerase. Proc Soc Exp Biol Med. 1997 Feb;214(2):99-106. doi: 10.3181/00379727-214-44075. PMID 9034126
- [Background] Sasaki M, Tanaka Y, Kaneuchi M, Sakuragi N, Dahiya R. CYP1B1 gene polymorphisms have higher risk for endometrial cancer, and positive correlations with estrogen receptor alpha and estrogen receptor beta expressions. Cancer Res. 2003 Jul 15;63(14):3913-8. PMID 12873984
- [Background] Kasperczyk H, La Ferla-Bruhl K, Westhoff MA, Behrend L, Zwacka RM, Debatin KM, Fulda S. Betulinic acid as new activator of NF-kappaB: molecular mechanisms and implications for cancer therapy. Oncogene. 2005 Oct 20;24(46):6945-56. doi: 10.1038/sj.onc.1208842. PMID 16007147
- [Background] Harley CB. Telomerase and cancer therapeutics. Nat Rev Cancer. 2008 Mar;8(3):167-79. doi: 10.1038/nrc2275. PMID 18256617
- [Background] Gollwitzer H, von Eisenhart-Rothe R, Holzapfel BM, Gradinger R. [Revision arthroplasty of the hip: acetabular component]. Chirurg. 2010 Apr;81(4):284-92. doi: 10.1007/s00104-009-1845-2. German. PMID 20232028
- [Background] Seydel C. Spotlight Therapeutics: making CRISPR deliver in vivo. Nat Biotechnol. 2021 Jul 14. doi: 10.1038/d41587-021-00011-9. Online ahead of print. No abstract available. PMID 34262172
- [Background] Uwe Platzbecker, Steven W Lane, Alice Garnier, Thomas Cluzeau, Odile Rauzy, Katharina S. S. Götze, Aristoteles Giagounidis, Deepak Singhal, Aicha Kopecky, Fatiha Chermat, Lionel Ades; A Phase II Study Evaluating the Efficacy and Safety of Imetelstat in Patients with Advanced Myelodysplastic Neoplasms or AML Failing HMA-Based Therapy - Interim Analysis Results of the Impress Study. Blood 2024; 144 (Supplement 1): 3222. doi: https://doi.org/10.1182/blood-2024-194185
- [Background] "Back Matter." Biometrics, vol. 14, no. 2, 1958. JSTOR, http://www.jstor.org/stable/2527794. Accessed 25 Nov. 2025.
- [Background] Brookmeyer, R., & Crowley, J. (1982). A Confidence Interval for the Median Survival Time. Biometrics, 38(1), 29-41. https://doi.org/10.2307/2530286